CLINICAL TRIAL: NCT01887821
Title: A Randomised Controlled Trial to Assess the Antimalarial Drug Susceptibility and Molecular Characterization of Plasmodium Vivax Isolates in Vietnam
Brief Title: Antimalarial Drug Susceptibility and Molecular Characterization of Plasmodium Vivax Isolates in Vietnam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Institute of Malaria, Parasitology and Entomology, Ho Chi Minh City, Viet Nam (Unknown); Hospital for Tropical Diseases, Ho Chi Minh City, Vietnam (Other); Agency for Science, Technology and Research (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07MA
Record Dates: First submitted 2013-06-19; First posted 2013-06-27 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2014-06

CONDITIONS: Plasmodium Vivax Malaria
MeSH Terms: conditions — Malaria, Vivax | interventions — Chloroquine; artenimol; piperaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroquine (Active Comparator): 25mg base/kg for 3 days
  Interventions: Drug: Chloroquine
- Dihydroartemisinin/Piperaquine (Active Comparator): Dihydroartemisinin 40 mg + piperaquine phosphate 320 mg per tablet; once daily for three days, doses depend on weight
  Interventions: Drug: Dihydroartemisinin/Piperaquine

INTERVENTIONS:
Drug: Chloroquine
  Arms: Chloroquine
Drug: Dihydroartemisinin/Piperaquine
  Arms: Dihydroartemisinin/Piperaquine

SUMMARY:
This is a study of drug effectiveness for 2 treatments of vivax malaria, which is one of the two main types of malaria in Viet Nam. There are two important drugs used in Viet Nam for treating vivax malaria, Chloroquine and Artemisinin. Sometimes, when medicines are used for many years they become less effective at treating a disease, especially when they are not used at adequate doses according to national guidelines or when counterfeit drugs are available in the market. The purpose of this study is to check that Chloroquine and Artemisinin, are still effective for patients in Viet Nam.

Participants in this study will be treated with either Dihydroartemisinin-Piperaquine (DHA-PPQ) or Chloroquine (CQ) for 3 days. Both drugs are recommended by the national guidelines to treat vivax malaria. The investigators would like to know if both of these treatments are equally effective so half of the patients in the study will be treated with DHA-PPQ and the other half will be treated with CQ. This way the investigators can compare the drugs to find out if one is better than the other.

Participants will be followed for 3 days in hospital, then regularly by follow-up visits until the 63rd day. Tests will be done to determine the amount of drug and malaria parasites in the participant's body and how the blood cells react to the malaria. The parasite will be tested to determine what type it is and how it reacts to the treatment.

The results of the study will be used to inform malaria treatment guidelines in Viet Nam.

ELIGIBILITY:
Inclusion Criteria:

* Age > 3 years;
* Mono-infection with P. vivax, parasitemia > 250/µl asexual forms for in vivo and >8000 asexual parasites/µl blood for in vitro testing;
* Presence of axillary or tympanic temperature ≥ 37.5 °C or history of fever during the past 24 h;
* Ability to swallow oral medication;
* Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule;
* Informed consent/assent

Exclusion Criteria:

* Presence of general danger signs or severe malaria according to the definitions of WHO (2000);
* Mixed infection with P.falciparum and P.vivax of other plasmodium species;
* Presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* Regular medication, which may interfere with antimalarial pharmacokinetics;
* Received antimalarial drugs in the previous 48 hours;
* History of hypersensitivity reactions or contraindications to any of the medicine(s) being tested or used as alternative treatment(s);
* Splenectomy;
* First trimester of pregnancy.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2013-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with adequate response to treatment | Day 63
  Adequate response = adequate clinical and parasitological response. Absence of parasitaemia on day 63, irrespective of temperature, in patients who did not previously meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure.

SECONDARY OUTCOMES:
Proportion of patients classified as Early Treatment Failures | Day 63
  One or more of the following:
  * danger signs or severe malaria on day 1, 2 or 3 in the presence of parasitaemia;
  * parasitaemia on day 2 higher than on day 0, irrespective of temperature;
  * parasitaemia on day 3 with temperature ≥ 37.5 ºC;
  * parasitaemia on day 3 ≥ 25% of count on day 0.
The parasite clearance time | Assessed every 6 hours until Day 3, or two consecutive parasite negative slides.
  Defined as the time in hours from the first treatment dose to the first of two consecutive parasitemia counts of zero.
Fever clearance time | Assessed every 6 hours until Day 3, or 24 hours without fever
  Defined as the time in hours from the first treatment dose to the start of the first sustained period of 24 hours without fever
Frequency of adverse and serious adverse events | Day 63
Proportion of patients classified as Late Clinical Failures | Day 63
  One or more of the following:
  * danger signs or severe malaria in the presence of parasitaemia on any day between day 4 and day 63 in patients who did not previously meet any of the criteria of early treatment failure;
  * presence of parasitaemia on any day between day 4 and day 63 with temperature ≥ 37.5 ºC (or history of fever) in patients who did not previously meet any of the criteria of early treatment failure
Proportion of patients classified as Late Parasitological Failures | Day 63
  Presence of parasitaemia on any day between day 7 and day 63 with temperature < 37.5 ºC in patients who did not previously meet any of the criteria of early treatment failure or late clinical failure

CONTACTS AND LOCATIONS:
Locations (1):
- Bu Gia Map Health Station, Phước Hòa, Binh Phuoc, Vietnam

REFERENCES:
- See also: Oxford University Clinical Research Unit, Viet Nam — http://www.oucru.org